CLINICAL TRIAL: NCT00780455
Title: Multicenter, Open Label, Randomized and Parallel Group Phase IV Pilot Study Evaluating the Effectiveness of Functional Rehabilitation Protocol in RRMS Patients Treated With Betaferon®
Brief Title: Rehabilitation Study in MS Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13089; 2006-006673-24 (EudraCT Number); 308083 (Other: Company internal)
Record Dates: First submitted 2008-05-28; First posted 2008-10-27 (Estimated); Results first posted 2013-02-26 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: KineSEP; Rehabilitation; Betaferon
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Interferon beta-1b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interferon beta-1b, FRP within 15 days after randomization (Experimental): Interferon beta-1b (Betaseron, BAY86-5046) 250 microgram (8 MUI), sub-cutaneous, administration every other day, Participants starting the 6 weeks functional rehabilitation protocol (FRP) within 15 days after randomization
  Interventions: Drug: Interferon beta-1b, FRP within 15 days after randomization
- Interferon beta-1b, FRP about 6 weeks after randomization (Experimental): Interferon beta-1b (Betaseron, BAY86-5046) 250 microgram (8 MUI), sub-cutaneous, administration every other day, Participants starting the 6 weeks functional rehabilitation protocol (FRP) about 6 weeks after randomization
  Interventions: Drug: Interferon beta-1b, FRP about 6 weeks after randomization

INTERVENTIONS:
Drug: Interferon beta-1b, FRP within 15 days after randomization — Treatment by Interferon beta-1b (Betaseron, BAY86-5046) for 3 month and beginning of the Functional Rehabilitation Program starting within 6 weeks after randomization
  Arms: Interferon beta-1b, FRP within 15 days after randomization
Drug: Interferon beta-1b, FRP about 6 weeks after randomization — Treatment by Interferon beta-1b (Betaseron, BAY86-5046) for 3 month and beginning of the Functional Rehabilitation Program about 6 weeks after randomization.
  Arms: Interferon beta-1b, FRP about 6 weeks after randomization

SUMMARY:
Studying the effectiveness of a functional rehabilitation protocol (FRP) in early Relapsing Remitting Multiple Sclerosis (RRMS) patients treated with Betaferon by comparing the physical ability of patients with and without FRP.

ELIGIBILITY:
Inclusion Criteria:

* Female and Male patients aged 18 and more;
* Confirmed diagnosis of RRMS according to the MacDonald or Poser criteria;
* First indication for Betaferon treatment (as described in Summary of Product Characteristics (SmPC));
* No relapse of multiple sclerosis (MS) in the last two months before the inclusion;
* Walking patients having an Expanded Disability Status Scale (EDSS) score between > 1 and </= 4 at the inclusion visit;
* Female of child-bearing potential must agree to practice adequate contraception methods over all the duration of the study;
* Patient can follow all the study and comply with all procedures of the trial protocol
* Laboratory evaluations (i.e. evaluation of hepatic enzymes gammaGT, full blood count and differential white blood cell [WBC]) must be available and the results must be normal;
* Written informed consent.

Exclusion Criteria:

* Any contraindication to Betaferon as described in the SmPC of the product;
* Patient with a previously orthopaedic surgical intervention within the past year of the inclusion;
* Patient previously included in this study;
* Patient previously treated within the past 3 months with Rebif, Avonex or Copaxone;
* Patient previously treated within the past 12 months with Betaferon;
* Participation in any clinical trial within the past 30 days involving the investigational drug intake.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (10):
- France (10):
  - Rennes, Brittany Region
  - Avignon
  - Lille
  - Lomme
  - Montpellier
  - Mulhouse
  - Nîmes
  - Quimper
  - Reims
  - Toulouse

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only 4 patients enrolled / 70 patients planned. Study stopped prematurely
Groups:
- Interferon Beta-1b, FRP Within 15 Days After Randomization: Interferon beta-1b (Betaseron, BAY86-5046) 250 microgram (8 MUI), sub-cutaneous, administration every other day, Participants starting the 6 weeks functional rehabilitation protocol (FRP) within 15 days after randomization. The FRP consisted of an intensive program over 6 weeks of effort and muscular reinforcement rehabilitation.
- Interferon Beta-1b, FRP About 6 Weeks After Randomization: Interferon beta-1b (Betaseron, BAY86-5046) 250 microgram (8 MUI), sub-cutaneous, administration every other day, Participants starting the 6 weeks functional rehabilitation protocol (FRP) about 6 weeks after randomization. The FRP consisted of an intensive program over 6 weeks of effort and muscular reinforcement rehabilitation.
Period: Overall Study
Arm/Group | Interferon Beta-1b, FRP Within 15 Days After Randomization | Interferon Beta-1b, FRP About 6 Weeks After Randomization
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interferon Beta-1b, FRP Within 15 Days After Randomization | Interferon Beta-1b, FRP About 6 Weeks After Randomization | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (16.3) | 45 (15.6) | 42.3 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Total Walking Area (in Covered Meters) Either After 6 Minute or at the Time of the Premature Stop of the Test.
Time Frame: Up to 6 minutes
Population: Due to the very low number of patients enrolled in the study, no statistical report was done.
Arm/Group | Interferon Beta-1b, FRP Within 15 Days After Randomization | Interferon Beta-1b, FRP About 6 Weeks After Randomization
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Time of Discomfort Appearance
Time Frame: Up to 6 minutes
Population: Due to the very low number of patients enrolled in the study, no statistical report was done.
Arm/Group | Interferon Beta-1b, FRP Within 15 Days After Randomization | Interferon Beta-1b, FRP About 6 Weeks After Randomization
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Distance of Discomfort Appearance
Time Frame: Up to 6 minutes
Population: Due to the very low number of patients enrolled in the study, no statistical report was done.
Arm/Group | Interferon Beta-1b, FRP Within 15 Days After Randomization | Interferon Beta-1b, FRP About 6 Weeks After Randomization
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Rhythm Change During 6 Minutes Walking Test
Time Frame: Up to 6 minutes
Population: Due to the very low number of patients enrolled in the study, no statistical report was done.
Arm/Group | Interferon Beta-1b, FRP Within 15 Days After Randomization | Interferon Beta-1b, FRP About 6 Weeks After Randomization
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Covered Distance Gain Between MR2 Visit and MR3 Visit
Description: Participants had the following two types of visit during the study, one visit with a neurologist and one visit with a rehabilitation physician. Visit to a neurologist: V0=baseline; V1=end of Month 1 of treatment; V2=end of Month 2 of treatment; V3=end of Month 3 of treatment. Visit to MR (Medecin Reeducateur: physician for rehabilitation): MR1=1st visit within 15 days after V0; MR2=2nd visit (6 weeks after MR1 +/- 1 week); MR3=end of study visit 12 weeks after MR1. This outcome was only measured on patients in the group "Interferon beta-1b, FRP within 15 days after randomization".
Time Frame: At MR2 visit (6 weeks after MR1 visit) and MR3 visit (12 weeks after MR1 visit)
Population: Due to the very low number of patients enrolled in the study, no statistical report was done.
Arm/Group | Interferon Beta-1b, FRP Within 15 Days After Randomization | Interferon Beta-1b, FRP About 6 Weeks After Randomization
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Knee Isokinetic Gain Between Baseline and 12 Weeks After MR1 Visit
Description: The isokinetic evaluation analyses the flexor/extensor ratio at different rates. The evaluation will be done at the beginning on the best clinical side otherwise on the strongest. Participants had the following two types of visit during the study, one visit with a neurologist and one visit with a rehabilitation physician. Visit to a neurologist: V0=baseline; V1=end of Month 1 of treatment; V2=end of Month 2 of treatment; V3=end of Month 3 of treatment. Visit to MR (Medecin Reeducateur: physician for rehabilitation): MR1=1st visit within 15 days after V0; MR2=2nd visit (6 weeks after MR1 +/- 1 week); MR3=end of study visit 12 weeks after MR1.
Time Frame: At baseline and 12 weeks after MR1 visit
Population: Due to the very low number of patients enrolled in the study, no statistical report was done.
Arm/Group | Interferon Beta-1b, FRP Within 15 Days After Randomization | Interferon Beta-1b, FRP About 6 Weeks After Randomization
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Posturography Gain in Static Equilibrium Performances Between Baseline and 12 Weeks After MR1 Visit
Description: Posturography protocol: Static equilibrium performances are evaluated in the standing patient on a fixed platform, in the standardized position (arms dangling, feet open at 30° and malleolus at a 5 cm distance). Participants had the following two types of visit during the study, one visit with a neurologist and one visit with a rehabilitation physician. Visit to a neurologist: V0=baseline; V1=end of Month 1 of treatment; V2=end of Month 2 of treatment; V3=end of Month 3 of treatment. Visit to MR (Medecin Reeducateur: physician for rehabilitation): MR1=1st visit within 15 days after V0; MR2=2nd visit (6 weeks after MR1 +/- 1 week); MR3=end of study visit 12 weeks after MR1.
Time Frame: At baseline and 12 weeks after MR1 visit
Population: Due to the very low number of patients enrolled in the study, no statistical report was done.
Arm/Group | Interferon Beta-1b, FRP Within 15 Days After Randomization | Interferon Beta-1b, FRP About 6 Weeks After Randomization
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Posturography Gain in Static Equilibrium Performances Between MR2 and MR3 Visits
Description: Posturography protocol: Static equilibrium performances are evaluated in the standing patient on a fixed platform, in the standardized position (arms dangling, feet open at 30° and malleolus at a 5 cm distance). Participants had the following two types of visit during the study, one visit with a neurologist and one visit with a rehabilitation physician. Visit to a neurologist: V0=baseline; V1=end of Month 1 of treatment; V2=end of Month 2 of treatment; V3=end of Month 3 of treatment. Visit to MR (Medecin Reeducateur: physician for rehabilitation): MR1=1st visit within 15 days after V0; MR2=2nd visit (6 weeks after MR1 +/- 1 week); MR3=end of study visit 12 weeks after MR1. This outcome was only measured on patients in the group "Interferon beta-1b, FRP within 15 days after randomization".
Time Frame: At MR2 visit (6 weeks after MR1 visit) and MR3 visit (12 weeks after MR1 visit)
Population: Due to the very low number of patients enrolled in the study, no statistical report was done.
Arm/Group | Interferon Beta-1b, FRP Within 15 Days After Randomization | Interferon Beta-1b, FRP About 6 Weeks After Randomization
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Participants With Fatigue Based on Participants Self Assessment Using the Fatigue Severity Scale (FSS)
Description: FSS is an auto-questionnaire estimating the fatigue. It includes 9 questions on 7 points as well as an analogical visual scale estimating the state of fatigue over the last two weeks. Participants had the following two types of visit during the study, one visit with a neurologist and one visit with a rehabilitation physician. Visit to a neurologist: V0=baseline; V1=end of Month 1 of treatment; V2=end of Month 2 of treatment; V3=end of Month 3 of treatment. Visit to MR (Medecin Reeducateur: physician for rehabilitation): MR1=1st visit within 15 days after V0; MR2=2nd visit (6 weeks after MR1 +/- 1 week); MR3=end of study visit 12 weeks after MR1.
Time Frame: From baseline to 12 weeks after MR1 visit
Population: Due to the very low number of patients enrolled in the study, no statistical report was done.
Arm/Group | Interferon Beta-1b, FRP Within 15 Days After Randomization | Interferon Beta-1b, FRP About 6 Weeks After Randomization
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Quality of Life Assessed by Use of Self-questionnaire (SEP-59)
Description: SEP (Sclérose en plaques) - 59: auto-questionnaire, multidimensional investigating the felt health. It contains a generic part SF (Short Form) 36 constituted by 36 items including the main concepts of quality of life and a specific part to the MS which investigates the dimensions susceptible to be degraded. 59 items are grouped in 16 dimensions: physical activity, limitations bound connected to the physical health, to the mental health, the social well-being, the pain, the energy, the emotional well-being, general Health, distress, cognitive function sexual function/satisfaction, well-being general, sleep and social support. Visit to a neurologist: V0=baseline; V1=end of Month 1 of treatment; V2=end of Month 2 of treatment; V3=end of Month 3 of treatment. Visit to MR (Medecin Reeducateur: physician for rehabilitation): MR1=1st visit within 15 days after V0; MR2=2nd visit (6 weeks after MR1 +/- 1 week); MR3=end of study visit 12 weeks after MR1.
Time Frame: From baseline to 12 weeks after MR1 visit
Population: Due to the very low number of patients enrolled in the study, no statistical report was done.
Arm/Group | Interferon Beta-1b, FRP Within 15 Days After Randomization | Interferon Beta-1b, FRP About 6 Weeks After Randomization
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Interferon Beta-1b, FRP Within 15 Days After Randomization | Interferon Beta-1b, FRP About 6 Weeks After Randomization
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interferon Beta-1b, FRP Within 15 Days After Randomization (N=2) | Interferon Beta-1b, FRP About 6 Weeks After Randomization (N=2)
Fatigue (General disorders) | 1 (1) | 1 (1)
Otitis external ear (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Mood trouble (Psychiatric disorders) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1) — transaminases increase
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0)
Urinary tract infections (Infections and infestations) | 0 (0) | 1 (1)
Tooth Extraction (General disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to the very low number of patients enrolled in the study, no statistical report was done. Study was early terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No